CLINICAL TRIAL: NCT01704287
Title: Randomized, Phase II Study of Pembrolizumab (MK-3475) Versus Chemotherapy in Patients With Advanced Melanoma (KEYNOTE 002)
Brief Title: Study of Pembrolizumab (MK-3475) Versus Chemotherapy in Participants With Advanced Melanoma (MK-3475-002/P08719/KEYNOTE-002)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P08719; MK-3475-002 (Other: Merck); 2012-003030-17 (EudraCT Number); KEYNOTE-002 (Other: Merck); P08719 (Other: Schering Plough)
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-04

CONDITIONS: Malignant Melanoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Carboplatin; Paclitaxel; Dacarbazine; Temozolomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Pembrolizumab 2 mg/kg (Experimental): Participants were initially randomized to receive pembrolizumab 2 mg/kg intravenously (IV) once every 3 weeks (Q3W). With Amendment 03, this dosing was discontinued and all study participants were to be treated with fixed-dose open label pembrolizumab 200 mg IV Q3W. Participants were to receive study drug until discontinuation due to progression of disease, toxicity, or choice. (Up to ~66 months)
  Interventions: Biological: Pembrolizumab
- Pembrolizumab 10 mg/kg (Experimental): Participants were initially randomized to receive pembrolizumab 10 mg/kg IV Q3W. With Amendment 03, this dosing was discontinued and all study participants were to be treated with fixed-dose open label pembrolizumab 200 mg IV Q3W. Participants were to receive study drug until discontinuation due to progression of disease, toxicity, or choice. (Up to ~66 months)
  Interventions: Biological: Pembrolizumab
- Investigator-Choice Chemotherapy (ICC) (Active Comparator): Participants were initially randomized to receive 1 of 4 possible chemotherapy regimens decided at the treating institution (carboplatin+paclitaxel, paclitaxel alone, dacarbazine, or temozolomide). Participants were to receive study drug until discontinuation due to progression of disease, toxicity, or choice. (Up to ~66 months)
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Dacarbazine; Drug: Temozolomide
- ICC→Pembrolizumab 2 mg/kg (Experimental): Participants who were initially randomized to ICC, subsequently experienced confirmed progressive disease (PD) and met all switching criteria at study treatment Week 12, had the opportunity to switch to receive pembrolizumab 2 mg/kg or 10 mg/kg. Participants received pembrolizumab 2 mg/kg IV Q3W. With Amendment 03, this dosing was discontinued and all study participants were to be treated with fixed-dose open label pembrolizumab 200 mg IV Q3W. Participants were to receive study drug until discontinuation due to PD, toxicity, or choice. (Up to ~66 months)
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Dacarbazine; Drug: Temozolomide
- ICC→Pembrolizumab 10 mg/kg (Experimental): Participants who were initially randomized to ICC, subsequently experienced confirmed progressive disease (PD) and met all switching criteria at study treatment Week 12, had the opportunity to switch to receive pembrolizumab 2 mg/kg or 10 mg/kg. Participants received pembrolizumab 10 mg/kg IV Q3W. With Amendment 03, this dosing was discontinued and all study participants were to be treated with fixed-dose open label pembrolizumab 200 mg IV Q3W. Participants were to receive study drug until discontinuation due to PD, toxicity, or choice. (Up to ~66 months)
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Dacarbazine; Drug: Temozolomide

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: SCH 900475; MK-3475; KEYTRUDA®
  Arms: ICC→Pembrolizumab 10 mg/kg; ICC→Pembrolizumab 2 mg/kg; Pembrolizumab 10 mg/kg; Pembrolizumab 2 mg/kg
Drug: Carboplatin — Carboplatin per institutional standard
  Other Names: PARAPLATIN®
  Arms: ICC→Pembrolizumab 10 mg/kg; ICC→Pembrolizumab 2 mg/kg; Investigator-Choice Chemotherapy (ICC)
Drug: Paclitaxel — Paclitaxel per institutional standard
  Other Names: TAXOL®
  Arms: ICC→Pembrolizumab 10 mg/kg; ICC→Pembrolizumab 2 mg/kg; Investigator-Choice Chemotherapy (ICC)
Drug: Dacarbazine — Dacarbazine per institutional standard
  Other Names: DTIC
  Arms: ICC→Pembrolizumab 10 mg/kg; ICC→Pembrolizumab 2 mg/kg; Investigator-Choice Chemotherapy (ICC)
Drug: Temozolomide — Temozolomide per institutional standard
  Other Names: TEMODAR®
  Arms: ICC→Pembrolizumab 10 mg/kg; ICC→Pembrolizumab 2 mg/kg; Investigator-Choice Chemotherapy (ICC)

SUMMARY:
This study was conducted to compare survival using pembrolizumab (SCH 900475, MK-3475) or standard chemotherapy in participants with advanced melanoma (MEL) who had progressed after prior therapy.

Initial Treatment Period:

Participants were initially randomized to receive either low-dose (2 mg/kg) pembrolizumab, higher dose (10 mg/kg) pembrolizumab or Investigator-choice chemotherapy (ICC). The four standard chemotherapy choices were: carboplatin + paclitaxel, paclitaxel alone, dacarbazine, or temozolomide. The randomization to either pembrolizumab or ICC was conducted in an open-label fashion.

The starting pembrolizumab dose was initially blinded to Investigators and participants until Amendment 03. With Amendment 03, all ongoing pembrolizumab participants were to be treated with open label, fixed dose pembrolizumab 200 mg, instead of a weight-based dosing of pembrolizumab.

Switch-to-Pembrolizumab Treatment Period:

Participants who were initially randomized to receive ICC and experienced progressive disease (PD) may have been eligible to switch to receiving pembrolizumab provided they met protocol-specified requirements for switching. Qualified participants were re-randomized to receive either pembrolizumab 2 mg/kg or pembrolizumab 10 mg/kg in a double-blind fashion. Participants who qualified to switch to pembrolizumab must have completed a washout period of ≥28 days from last dose of chemotherapy before receiving pembrolizumab. With Amendment 03, all switched-to-pembrolizumab participants were to be treated with open-label, fixed dose pembrolizumab 200 mg instead of a weight-based dosing of pembrolizumab.

DETAILED DESCRIPTION:
Two interim and one final statistical analyses were planned for and conducted during this study:

* Interim Analysis 1 (futility analysis),
* Interim Analysis 2 (~18 months into study): database cutoff date 12-May-2014, and
* Final Analysis (~36 months into study): database cutoff date 16-Nov-2015. The End of Trial Analysis for the study was conducted at ~75 months into the study: database cutoff date 31-Jan-2019.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of unresectable Stage III or metastatic MEL not amenable to local therapy
* Participants must be refractory to ipilimumab
* Participants with BRAF gene mutant melanoma must have had a prior treatment regimen that included vemurafenib, dabrafenib, or an approved BRAF gene and/or mitogen-activated protein kinase (MEK) protein inhibitor
* Must consent to allow correlative studies; must provide a newly obtained tissue/biopsy specimen (or specimen obtained within 60 days of consenting)
* Radiographically measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Chemotherapy, radiation therapy, or biological cancer therapy within 4 weeks prior to the first dose of study drug, or not recovered from the AEs due to cancer therapies administered more than 4 weeks earlier
* Disease progression within 24 weeks of last dose of ipilimumab
* Participating or has participated in a study of an investigational agent or using an investigational device within 30 days of the first dose of study drug
* Expected to require any other form of systemic or localized antineoplastic therapy while on study
* Chronic systemic steroid therapy within 2 weeks before the planned date for first dose randomized treatment or on any other form of immunosuppressive medication
* Known history of any other than the current malignancy excepting adequately treated basal or squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, breast cancer, or other in situ cancers
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active autoimmune disease or a history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents
* Prior treatment with any other anti-programmed cell death (PD) agent
* Active infection requiring systemic therapy
* Known history of Human Immunodeficiency Virus (HIV)
* Active Hepatitis B or Hepatitis C
* Regular user (including recreational use of) illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol)
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study through 120 days after last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2012-11-20 (Actual); Primary Completion 2015-11-16 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Ribas A, Puzanov I, Dummer R, Schadendorf D, Hamid O, Robert C, Hodi FS, Schachter J, Pavlick AC, Lewis KD, Cranmer LD, Blank CU, O'Day SJ, Ascierto PA, Salama AK, Margolin KA, Loquai C, Eigentler TK, Gangadhar TC, Carlino MS, Agarwala SS, Moschos SJ, Sosman JA, Goldinger SM, Shapira-Frommer R, Gonzalez R, Kirkwood JM, Wolchok JD, Eggermont A, Li XN, Zhou W, Zernhelt AM, Lis J, Ebbinghaus S, Kang SP, Daud A. Pembrolizumab versus investigator-choice chemotherapy for ipilimumab-refractory melanoma (KEYNOTE-002): a randomised, controlled, phase 2 trial. Lancet Oncol. 2015 Aug;16(8):908-18. doi: 10.1016/S1470-2045(15)00083-2. Epub 2015 Jun 23. PMID 26115796
- [Result] Hamid O, Puzanov I, Dummer R, Schachter J, Daud A, Schadendorf D, Blank C, Cranmer LD, Robert C, Pavlick AC, Gonzalez R, Hodi FS, Ascierto PA, Salama AKS, Margolin KA, Gangadhar TC, Wei Z, Ebbinghaus S, Ibrahim N, Ribas A. Final analysis of a randomised trial comparing pembrolizumab versus investigator-choice chemotherapy for ipilimumab-refractory advanced melanoma. Eur J Cancer. 2017 Nov;86:37-45. doi: 10.1016/j.ejca.2017.07.022. PMID 28961465
- [Derived] Cristescu R, Aurora-Garg D, Albright A, Xu L, Liu XQ, Loboda A, Lang L, Jin F, Rubin EH, Snyder A, Lunceford J. Tumor mutational burden predicts the efficacy of pembrolizumab monotherapy: a pan-tumor retrospective analysis of participants with advanced solid tumors. J Immunother Cancer. 2022 Jan;10(1):e003091. doi: 10.1136/jitc-2021-003091. PMID 35101941
- [Derived] Robert C, Hwu WJ, Hamid O, Ribas A, Weber JS, Daud AI, Hodi FS, Wolchok JD, Mitchell TC, Hersey P, Dronca R, Joseph RW, Boutros C, Min L, Long GV, Schachter J, Puzanov I, Dummer R, Lin J, Ibrahim N, Diede SJ, Carlino MS, Joshua AM. Long-term safety of pembrolizumab monotherapy and relationship with clinical outcome: A landmark analysis in patients with advanced melanoma. Eur J Cancer. 2021 Feb;144:182-191. doi: 10.1016/j.ejca.2020.11.010. Epub 2020 Dec 24. PMID 33360855
- [Derived] Lala M, Li TR, de Alwis DP, Sinha V, Mayawala K, Yamamoto N, Siu LL, Chartash E, Aboshady H, Jain L. A six-weekly dosing schedule for pembrolizumab in patients with cancer based on evaluation using modelling and simulation. Eur J Cancer. 2020 May;131:68-75. doi: 10.1016/j.ejca.2020.02.016. Epub 2020 Apr 15. PMID 32305010
- [Derived] van Vugt MJH, Stone JA, De Greef RHJMM, Snyder ES, Lipka L, Turner DC, Chain A, Lala M, Li M, Robey SH, Kondic AG, De Alwis D, Mayawala K, Jain L, Freshwater T. Immunogenicity of pembrolizumab in patients with advanced tumors. J Immunother Cancer. 2019 Aug 8;7(1):212. doi: 10.1186/s40425-019-0663-4. PMID 31395089
- [Derived] Wang M, Chen C, Jemielita T, Anderson J, Li XN, Hu C, Kang SP, Ibrahim N, Ebbinghaus S. Are tumor size changes predictive of survival for checkpoint blockade based immunotherapy in metastatic melanoma? J Immunother Cancer. 2019 Feb 8;7(1):39. doi: 10.1186/s40425-019-0513-4. PMID 30736858
- [Derived] Hamid O, Robert C, Ribas A, Hodi FS, Walpole E, Daud A, Arance AS, Brown E, Hoeller C, Mortier L, Schachter J, Long J, Ebbinghaus S, Ibrahim N, Butler M. Antitumour activity of pembrolizumab in advanced mucosal melanoma: a post-hoc analysis of KEYNOTE-001, 002, 006. Br J Cancer. 2018 Sep;119(6):670-674. doi: 10.1038/s41416-018-0207-6. Epub 2018 Sep 11. PMID 30202085
- [Derived] Schadendorf D, Dummer R, Hauschild A, Robert C, Hamid O, Daud A, van den Eertwegh A, Cranmer L, O'Day S, Puzanov I, Schachter J, Blank C, Salama A, Loquai C, Mehnert JM, Hille D, Ebbinghaus S, Kang SP, Zhou W, Ribas A. Health-related quality of life in the randomised KEYNOTE-002 study of pembrolizumab versus chemotherapy in patients with ipilimumab-refractory melanoma. Eur J Cancer. 2016 Nov;67:46-54. doi: 10.1016/j.ejca.2016.07.018. Epub 2016 Sep 2. PMID 27596353
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This end of trial analysis is based on a trial closure database cutoff date of 31-Jan-2019.
Period: Initial Treatment Period
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Investigator-Choice Chemotherapy (ICC) | ICC→Pembrolizumab 2 mg/kg | ICC→Pembrolizumab 10 mg/kg
Started | 180 | 181 | 179 | 0 | 0
Treated | 178 | 179 | 171 | 0 | 0
Completed | 33 | 47 | 6 | 0 | 0
Not Completed | 147 | 134 | 173 | 0 | 0
Not completed — Death | 139 | 129 | 71 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 4 | 0 | 0
Not completed — Lost to Follow-up | 5 | 3 | 0 | 0 | 0
Not completed — Switched to Pembrolizumab | 0 | 0 | 98 | 0 | 0
Period: Switch to Pembrolizumab Treatment Period
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Investigator-Choice Chemotherapy (ICC) | ICC→Pembrolizumab 2 mg/kg | ICC→Pembrolizumab 10 mg/kg
Started | 0 | 0 | 0 | 53 | 45
Completed | 0 | 0 | 0 | 15 | 7
Not Completed | 0 | 0 | 0 | 38 | 38
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 1
Not completed — Death | 0 | 0 | 0 | 35 | 37
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consisted of all randomized participants. Participants were included in the group to which they were initially randomized for Baseline Characteristics.
Groups:
- Pembrolizumab 2 mg/kg: Participants were initially randomized to receive pembrolizumab 2 mg/kg IV Q3W. With Amendment 03, this dosing was discontinued and all study participants were to be treated with fixed-dose open label pembrolizumab 200 mg IV Q3W. Participants were to receive study drug until discontinuation due to progression of disease, toxicity, or choice. (Up to ~66 months)
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Investigator-Choice Chemotherapy (ICC) | Total
Number analyzed (Participants) | 180 | 181 | 179 | 540
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (14.9) | 60.1 (13.3) | 60.5 (12.7) | 60.1 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 72 | 65 | 213
  Male | 104 | 109 | 114 | 327
Programmed Cell Death-Ligand 1 (PD-L1) Tumor Expression Status [Count of Participants; unit: Participants] — Membranous PD-L1 expression in tumor and tumor-associated immune cells was assessed by immunohistochemistry assay and scored on a unique melanoma (Allred Proportion Score [APS]/Melanoma [MEL]) scale of 0 to 5 points. Participants with an APS score of ≥2 (membranous staining in ≥1% of cells) were considered to be PD-L1 Positive and participants with an APS score of 0 or 1 were considered to be PD-L1 Negative.
  Participants
    PD-L1 Positive | 99 | 97 | 98 | 294
    PD-L1 Negative | 48 | 46 | 40 | 134
    Unknown | 33 | 38 | 41 | 112

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) - Initial Treatment Period
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per Response Criteria in Solid Tumors version 1.1 (RECIST 1.1), PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions was also considered PD. Analysis of PFS was based on an integrated radiology and oncology (IRO) assessment and was not planned or conducted for the switch-to-pembrolizumab treatment groups. Median PFS based on the product limit (Kaplan-Meier) method for censored data is presented. This was the final analysis for PFS.
Time Frame: Up to approximately 36 months (Through Final Analysis database cutoff date of 16-Nov-2015)
Population: The analysis population consisted of all randomized participants. Participants were included in the initial treatment group to which they were randomized for the efficacy analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Investigator-Choice Chemotherapy (ICC)
Number analyzed (Participants) | 180 | 181 | 179
Months | 2.9 [2.8 to 3.8] | 3.0 [2.8 to 5.2] | 2.8 [2.6 to 2.8]
Statistical Analysis 1: Comparison: Pembrolizumab 2 mg/kg vs Investigator-Choice Chemotherapy (ICC); Test type: Superiority or Other — Cox regression model with treatment as covariate stratified by Eastern Cooperative Oncology Group (ECOG) performance status (0 vs. 1); lactate dehydrogenase (LDH) levels (normal vs. elevated LDH levels [≥110% Upper Limit of Normal (ULN)]); & BRAF mutational status (mutant vs. wild-type); p < 0.0001, Log Rank — One-sided p-value based on stratified log rank test; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.46 to 0.73] — Numerator=Pembrolizumab 2 mg/kg Denominator=ICC
Statistical Analysis 2: Comparison: Pembrolizumab 10 mg/kg vs Investigator-Choice Chemotherapy (ICC); Test type: Superiority or Other — Cox regression model with treatment as covariate stratified by ECOG performance status (0 vs. 1); LDH levels (normal vs. elevated LDH levels [≥110% ULN]); & BRAF mutational status (mutant vs. wild-type); p < 0.0001, Log Rank — One-sided p-value based on stratified log rank test; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.37 to 0.60] — Numerator=Pembrolizumab 10 mg/kg Denominator=ICC
Statistical Analysis 3: Comparison: Pembrolizumab 2 mg/kg vs Pembrolizumab 10 mg/kg; Test type: Superiority or Other — [test comment as in outcome 1, analysis 2]; p = 0.1247, Log Rank — Two-sided p-value based on stratified log rank test; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.66 to 1.05] — Numerator=Pembrolizumab 10 mg/kg Denominator=Pembrolizumab 2 mg/kg

2. Primary Outcome: Interim Overall Survival (OS) - Initial Treatment Period
Description: OS was defined as the time from randomization to death due to any cause. Analysis of OS was not planned or conducted for the switch-to-pembrolizumab treatment groups. Median OS based on the product-limit (Kaplan-Meier) method for censored data is presented. This was the interim analysis for OS.
Time Frame: Up to approximately 36 months (Through Final Analysis database cutoff date of 16-Nov-2015)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Investigator-Choice Chemotherapy (ICC)
Number analyzed (Participants) | 180 | 181 | 179
Months | 13.4 [11.0 to 16.4] | 14.7 [11.3 to 19.5] | 11.0 [8.9 to 13.8]
Statistical Analysis 1: Comparison: Pembrolizumab 2 mg/kg vs Investigator-Choice Chemotherapy (ICC); Cox regression model with treatment as covariate stratified by ECOG performance status (0 vs. 1); LDH levels (normal vs. elevated LDH levels [≥110% ULN]); & BRAF mutational status (mutant vs. wild-type); Test type: Superiority or Other; p = 0.1173, Log Rank — One-sided p-value based on stratified log rank test; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.67 to 1.10] — Numerator=Pembrolizumab 2 mg/kg Denominator=ICC
Statistical Analysis 2: Comparison: Pembrolizumab 10 mg/kg vs Investigator-Choice Chemotherapy (ICC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0106, Log Rank — One-sided p-value based on stratified log rank test; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.57 to 0.96] — Numerator=Pembrolizumab 10 mg/kg Denominator=ICC
Statistical Analysis 3: Comparison: Pembrolizumab 2 mg/kg vs Pembrolizumab 10 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2905, Log Rank — Two-sided p-value based on stratified log rank test; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.67 to 1.12] — Numerator=Pembrolizumab 10 mg/kg Denominator=Pembrolizumab 2 mg/kg

3. Primary Outcome: Final Overall Survival (OS) - Initial Treatment Period
Description: OS was defined as the time from randomization to death due to any cause. Analysis of OS was not planned or conducted for the switch-to-pembrolizumab treatment groups. Median OS duration based on the product-limit (Kaplan-Meier) method for censored data is presented. This was the final analysis for OS.
Time Frame: Up to approximately 75 months (Through End of Trial Analysis database cutoff date of 31-Jan-2019)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Investigator-Choice Chemotherapy (ICC)
Number analyzed (Participants) | 180 | 181 | 179
Months | 13.4 [11.0 to 16.4] | 14.7 [11.3 to 19.5] | 11.0 [8.9 to 13.8]
Statistical Analysis 1: Comparison: Pembrolizumab 2 mg/kg vs Investigator-Choice Chemotherapy (ICC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1146, Log Rank — One-sided p-value based on stratified log rank test; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.68 to 1.10] — Numerator=Pembrolizumab 2 mg/kg Denominator=ICC
Statistical Analysis 2: Comparison: Pembrolizumab 10 mg/kg vs Investigator-Choice Chemotherapy (ICC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0023, Log Rank — One-sided p-value based on stratified log rank test; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.55 to 0.90] — Numerator=Pembrolizumab 10 mg/kg Denominator=ICC
Statistical Analysis 3: Comparison: Pembrolizumab 2 mg/kg vs Pembrolizumab 10 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1490, Log Rank — Two-sided p-value based on stratified log rank test; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.66 to 1.07] — Numerator=Pembrolizumab 10 mg/kg Denominator=Pembrolizumab 2 mg/kg

4. Secondary Outcome: Final Overall Survival (OS) By Programmed Cell Death-Ligand 1 (PD-L1) Tumor Expression Status - Initial Treatment Period
Description: OS was defined as the time from randomization to death due to any cause. Participants with an Allred Proportion Score (APS) ≥2 (membranous staining in ≥1% of cells for PD-L1) were considered to be PD-L1 Positive and participants with an APS of 0 or 1 were considered to be PD-L1 Negative. Analysis of OS was not planned or conducted for the switch-to-pembrolizumab treatment groups. Median OS duration based on the product-limit (Kaplan-Meier) method for censored data by PD-L1 tumor expression status is presented.
Time Frame: Up to approximately 75 months (Through End of Trial Analysis database cutoff date of 31-Jan-2019)
Population: The analysis population consisted of all randomized participants who had a PD-L1 tumor expression status assessment. Participants were included in the initial treatment group to which they were randomized for the efficacy analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Investigator-Choice Chemotherapy (ICC)
Number analyzed (Participants) | 180 | 181 | 179
Months
  PD-L1 Positive: number analyzed (Participants) | 99 | 97 | 98
  PD-L1 Positive | 15.0 [10.9 to 20.9] | 17.5 [13.7 to 28.9] | 12.1 [7.7 to 18.2]
  PD-L1 Negative: number analyzed (Participants) | 48 | 46 | 40
  PD-L1 Negative | 10.5 [6.4 to 13.5] | 13.4 [4.6 to 23.3] | 9.3 [5.1 to 14.2]
Statistical Analysis 1: Comparison: Pembrolizumab 2 mg/kg vs Investigator-Choice Chemotherapy (ICC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other — PD-L1-Positive Participants; p = 0.3113, Log Rank — One-sided p-value based on stratified log rank test; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.66 to 1.28] — Numerator=Pembrolizumab 2 mg/kg Denominator=ICC
Statistical Analysis 2: Comparison: Pembrolizumab 10 mg/kg vs Investigator-Choice Chemotherapy (ICC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other — PD-L1 Positive Participants; p = 0.0208, Log Rank — One-sided p-value based on stratified log rank test; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.50 to 0.99] — Numerator=Pembrolizumab 10 mg/kg Denominator=ICC
Statistical Analysis 3: Comparison: Pembrolizumab 2 mg/kg vs Pembrolizumab 10 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other — PD-L1 Positive Participants; p = 0.0496, Log Rank — Two-sided p-value based on stratified log rank test; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.50 to 1.00] — Numerator=Pembrolizumab 10 mg/kg Denominator=Pembrolizumab 2 mg/kg
Statistical Analysis 4: Comparison: Pembrolizumab 2 mg/kg vs Investigator-Choice Chemotherapy (ICC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other — PD-L1 Negative Participants; p = 0.6043, Log Rank — One-sided p-value based on stratified log rank test; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.65 to 1.76] — Numerator=Pembrolizumab 2 mg/kg Denominator=ICC
Statistical Analysis 5: Comparison: Pembrolizumab 10 mg/kg vs Investigator-Choice Chemotherapy (ICC); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other — PD-L1 Negative Participants; p = 0.0335, Log Rank — One-sided p-value based on stratified log rank test; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.37 to 1.04] — Numerator=Pembrolizumab 10 mg/kg Denominator=ICC
Statistical Analysis 6: Comparison: Pembrolizumab 2 mg/kg vs Pembrolizumab 10 mg/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other — PD-L1 Negative Participants; p = 0.1504, Log Rank — Two-sided p-value based on stratified log rank test; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.44 to 1.13] — Numerator=Pembrolizumab 10 mg/kg Denominator=Pembrolizumab 2 mg/kg

5. Secondary Outcome: Overall Response Rate (ORR) - Initial Treatment Period
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed using RECIST 1.1. Analysis of ORR was not planned or conducted for the switch-to-pembrolizumab treatment groups. The percentage of participants who experienced a CR or PR is presented. This was the final analysis for ORR.
Time Frame: Up to approximately 36 months (Through Final Analysis database cutoff date of 16-Nov-2015)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Investigator-Choice Chemotherapy (ICC)
Number analyzed (Participants) | 180 | 181 | 179
Percentage of Participants | 22.2 [16.4 to 29.0] | 27.6 [21.3 to 34.7] | 4.5 [1.9 to 8.6]

6. Secondary Outcome: Best Overall Response (BOR) - Initial Treatment Period
Description: BOR was assessed by independent radiology review using RECIST 1.1 and was recorded from randomization until the last imaging assessment in this period. Response categories included: Complete Response (CR): disappearance of all target lesions; Partial Response (PR): at least a 30% decrease in the sum of diameters of target lesions; Progressive Disease (PD): at least a 20% increase in the sum of diameters of target lesions; and Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. BOR for the Initial Treatment Period was based on IRO. BOR for participants during the Initial Treatment Period is presented.
Time Frame: Up to approximately 36 months (Through Final Analysis database cutoff date of 16-Nov-2015)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Investigator-Choice Chemotherapy (ICC)
Number analyzed (Participants) | 180 | 181 | 179
Percentage of Participants
  Complete Response | 3.3 [16.4 to 29.0] | 7.2 [21.3 to 34.7] | 0.0 [1.9 to 8.6]
  Partial Response | 18.9 | 20.4 | 4.5
  Stable Disease | 16.7 | 14.9 | 19.0
  Progressive Disease | 46.7 | 47.5 | 61.5
  Not Evaluable | 13.3 | 9.9 | 15.1
  No Disease | 0.6 | 0.0 | 0.0
  No Assessment | 0.6 | 0.0 | 0.0

7. Secondary Outcome: Best Overall Response (BOR) - Switch-to-Pembrolizumab Treatment Period
Description: The BOR was assessed using RECIST 1.1 and was recorded from the start of the second line of study drug (pembrolizumab) until the last imaging assessment in this period. Response categories included: Complete Response (CR): disappearance of all target lesions; Partial Response (PR): at least a 30% decrease in the sum of diameters of target lesions; Progressive Disease (PD): at least a 20% increase in the sum of diameters of target lesions; and Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. For the switch-to-pembrolizumab treatment groups, BOR was based on independent review committee (IRC) assessment. The BOR for switched-to pembrolizumab treatment groups is presented.
Time Frame: Up to approximately 36 months (Through Final Analysis database cutoff date of 16-Nov-2015)
Population: The analysis population consisted of all randomized participants in ICC who switched to receiving pembrolizumab. Participants were included in the treatment group to which they were re-randomized (switched) for this efficacy analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | ICC→Pembrolizumab 2 mg/kg | ICC→Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 53 | 45
Percentage of Participants
  Complete Response | 1.9 | 4.4
  Partial Response | 17.0 | 13.3
  Stable Disease | 15.1 | 11.1
  Progressive Disease | 54.7 | 55.6
  Not Evaluable | 11.3 | 13.3
  No Assessment | 0.0 | 2.2

8. Secondary Outcome: Duration of Response (DOR) - Initial Treatment Period
Description: For participants who demonstrated a confirmed response (Complete Response [CR]: disappearance of all target lesions or Partial Response [PR]: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death. DOR for participants who had not progressed or died at the time of analysis was to be censored at the date of their last tumor assessment. DOR analysis was based on IRO assessment. Analysis of DOR was not planned or analyzed for the switch-to-pembrolizumab treatment groups. Median DOR for participants who demonstrated a confirmed response is presented.
Time Frame: Up to approximately 36 months (Through Final Analysis database cutoff date of 16-Nov-2015)
Population: The analysis population consisted of all randomized participants who demonstrated a confirmed response (CR or PR) per RECIST 1.1. Participants were included in the initial treatment group to which they were randomized for the efficacy analysis.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | Investigator-Choice Chemotherapy (ICC)
Number analyzed (Participants) | 40 | 50 | 8
Months | 22.8 [1.4 to 25.3] | NA [1.1 to NA] — NA=DOR Median not reached NA=DOR Upper Limit not reached: no progressive disease by time of last assessment | 6.8 [2.8 to 11.3]

9. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE) - Overall Study
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of study drug, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition which was temporally associated with the use of study drug, was also an AE. Participants were included in the treatment group in which an AE was experienced. The number of participants who experienced at least one AE is presented.
Time Frame: Up to approximately 75 months (Through End of Trial Analysis database cutoff date of 31-Jan-2019)
Population: The analysis population consisted of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- ICC Only: Participants were randomized to receive 1 of 4 possible chemotherapy regimens decided at the treating institution (carboplatin+paclitaxel, paclitaxel alone, dacarbazine, or temozolomide). This treatment group included the participants who remained on ICC through the database cutoff date. Participants were to receive study drug until discontinuation due to progression of disease, toxicity, or choice. (Up to ~66 months)
- ICC→Pembrolizumab 2 mg/kg (After Switch to Pembrolizumab): Participants who were initially randomized to ICC, subsequently experienced confirmed progressive disease (PD) and met all switching criteria at study treatment Week 12, had the opportunity to switch to receive pembrolizumab 2 mg/kg or 10 mg/kg. Participants received pembrolizumab 2 mg/kg IV Q3W. With Amendment 03, this dosing was discontinued and all study participants were to be treated with fixed-dose open label pembrolizumab 200 mg IV Q3W. Participants were to receive study drug until discontinuation due to PD, toxicity, or choice. (Up to ~66 months)
- ICC→Pembrolizumab 10 mg/kg (After Switch to Pembrolizumab): Participants who were initially randomized to ICC, subsequently experienced confirmed progressive disease (PD) and met all switching criteria at study treatment Week 12, had the opportunity to switch to receive pembrolizumab 2 mg/kg or 10 mg/kg. Participants received pembrolizumab 10 mg/kg IV Q3W. With Amendment 03, this dosing was discontinued and all study participants were to be treated with fixed-dose open label pembrolizumab 200 mg IV Q3W. Participants were to receive study drug until discontinuation due to PD, toxicity, or choice. (Up to ~66 months)
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | ICC Only | ICC→Pembrolizumab 2 mg/kg | ICC→Pembrolizumab 10 mg/kg | ICC→Pembrolizumab 2 mg/kg (After Switch to Pembrolizumab) | ICC→Pembrolizumab 10 mg/kg (After Switch to Pembrolizumab)
Number analyzed (Participants) | 178 | 179 | 73 | 53 | 45 | 53 | 45
Participants | 172 | 179 | 71 | 52 | 45 | 53 | 41

10. Secondary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event (AE) - Overall Study
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition which is temporally associated with the use of study drug, was also an AE. The number of participants who discontinued study drug due to an AE is presented.
Time Frame: Up to approximately 75 months (Through End of Trial Analysis database cutoff date of 31-Jan-2019)
Population: The analysis population consisted of all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | ICC Only | ICC→Pembrolizumab 2 mg/kg | ICC→Pembrolizumab 10 mg/kg | ICC→Pembrolizumab 2 mg/kg (After Switch to Pembrolizumab) | ICC→Pembrolizumab 10 mg/kg (After Switch to Pembrolizumab)
Number analyzed (Participants) | 178 | 179 | 73 | 53 | 45 | 53 | 45
Participants | 29 | 33 | 13 | 1 | 1 | 4 | 4

ADVERSE EVENTS:
Time Frame: Up to approximately 75 months (Through End of Trial Analysis database cutoff date of 31-Jan-2019)
Description: Safety Population: All participants who received ≥1 dose of study drug. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study drug. Therefore, Medical Dictionary for Regulatory Activities (MedDRA) preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Groups:
- Investigator-Choice Chemotherapy (ICC) Only: Participants received 1 of 4 possible chemotherapy regimens decided at the treating institution (carboplatin+paclitaxel, paclitaxel alone, dacarbazine, or temozolomide). This treatment group included the participants who remained on ICC through the final analysis. Participants were to receive study drug until discontinuation due to progression of disease, toxicity, or choice. (Up to ~66 months)
- ICC→Pembrolizumab 2 mg/kg (Before Switch to Pembrolizumab); ICC→Pembrolizumab 2 mg/kg (After Switch to Pembrolizumab): Participants who were initially randomized to ICC, subsequently experienced confirmed progressive disease (PD) and met all switching criteria at study treatment Week 12, had the opportunity to switch to receive pembrolizumab 2 mg/kg or 10 mg/kg. Participants received pembrolizumab 2 mg/kg IV Q3W. With Amendment 03, this dosing was discontinued and all study participants were to be treated with fixed-dose open label pembrolizumab 200 mg IV Q3W. Participants were to receive study drug until discontinuation due to PD, toxicity, or choice. (Up to ~66 months)
- ICC→Pembrolizumab 10 mg/kg (Before Switch to Pembrolizumab): Participants who were initially randomized to ICC, subsequently experienced confirmed progressive disease (PD) and met all switching criteria at study treatment Week 12, had the opportunity to switch to receive pembrolizumab 2 mg/kg or 10 mg/kg. Participants received pembrolizumab 10 mg/kg IV Q3W. With Amendment 03, this dosing was discontinued and all study participants were to be treated with fixed-dose open label pembrolizumab 200 mg IV Q3W. Participants were to receive study drug until discontinuation due to PD, toxicity, or choice. (Up to ~66 months)
- ICC→Pembrolizumab 10 mg/kg (After Switch to Pembrolizumab): Participants who were initiall randomized to ICC, subsequently experienced confirmed progressive disease (PD) and met all switching criteria at study treatment Week 12, had the opportunity to switch to receive pembrolizumab 2 mg/kg or 10 mg/kg. Participants received pembrolizumab 10 mg/kg IV Q3W. With Amendment 03, this dosing was discontinued and all study participants were to be treated with fixed-dose open label pembrolizumab 200 mg IV Q3W. Participants were to receive study drug until discontinuation due to PD, toxicity, or choice. (Up to ~66 months)
Arm/Group | Investigator-Choice Chemotherapy (ICC) Only | ICC→Pembrolizumab 2 mg/kg (Before Switch to Pembrolizumab) | ICC→Pembrolizumab 10 mg/kg (Before Switch to Pembrolizumab) | Pembrolizumab 2 mg/kg | Pembrolizumab 10 mg/kg | ICC→Pembrolizumab 2 mg/kg (After Switch to Pembrolizumab) | ICC→Pembrolizumab 10 mg/kg (After Switch to Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 71/73 | 0/53 | 0/45 | 139/178 | 129/179 | 35/53 | 37/45
Serious Adverse Events (participants affected / at risk) | 33/73 | 15/53 | 9/45 | 91/178 | 78/179 | 18/53 | 18/45
Other Adverse Events (participants affected / at risk) | 66/73 | 52/53 | 44/45 | 158/178 | 176/179 | 48/53 | 36/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigator-Choice Chemotherapy (ICC) Only (N=73) | ICC→Pembrolizumab 2 mg/kg (Before Switch to Pembrolizumab) (N=53) | ICC→Pembrolizumab 10 mg/kg (Before Switch to Pembrolizumab) (N=45) | Pembrolizumab 2 mg/kg (N=178) | Pembrolizumab 10 mg/kg (N=179) | ICC→Pembrolizumab 2 mg/kg (After Switch to Pembrolizumab) (N=53) | ICC→Pembrolizumab 10 mg/kg (After Switch to Pembrolizumab) (N=45)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 3 (5) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac ventricular disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Addison's disease (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye movement disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 4 (5) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatic necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiation necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis noninfective (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myasthenic syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poor venous access (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical spine stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigator-Choice Chemotherapy (ICC) Only (N=73) | ICC→Pembrolizumab 2 mg/kg (Before Switch to Pembrolizumab) (N=53) | ICC→Pembrolizumab 10 mg/kg (Before Switch to Pembrolizumab) (N=45) | Pembrolizumab 2 mg/kg (N=178) | Pembrolizumab 10 mg/kg (N=179) | ICC→Pembrolizumab 2 mg/kg (After Switch to Pembrolizumab) (N=53) | ICC→Pembrolizumab 10 mg/kg (After Switch to Pembrolizumab) (N=45)
Anaemia (Blood and lymphatic system disorders) | 21 (26) | 15 (25) | 10 (10) | 30 (43) | 26 (31) | 12 (13) | 8 (21)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 16 (17) | 15 (16) | 4 (4) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 8 (10) | 1 (2) | 4 (4) | 28 (38) | 27 (33) | 7 (7) | 2 (3)
Constipation (Gastrointestinal disorders) | 16 (19) | 12 (17) | 8 (10) | 40 (47) | 42 (57) | 12 (14) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 13 (20) | 11 (17) | 11 (17) | 40 (52) | 41 (67) | 16 (23) | 9 (22)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (3) | 3 (3) | 3 (3) | 4 (5) | 4 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 23 (30) | 29 (44) | 19 (23) | 44 (74) | 49 (56) | 12 (12) | 10 (17)
Vomiting (Gastrointestinal disorders) | 17 (22) | 10 (14) | 13 (14) | 19 (26) | 38 (58) | 6 (7) | 2 (2)
Asthenia (General disorders) | 10 (11) | 4 (4) | 2 (2) | 19 (25) | 20 (44) | 2 (2) | 3 (3)
Fatigue (General disorders) | 28 (34) | 27 (36) | 26 (33) | 74 (106) | 91 (117) | 15 (17) | 16 (24)
Influenza like illness (General disorders) | 1 (2) | 1 (1) | 1 (1) | 9 (13) | 14 (17) | 4 (4) | 3 (6)
Oedema peripheral (General disorders) | 4 (4) | 5 (5) | 1 (1) | 17 (19) | 21 (24) | 6 (7) | 2 (2)
Pain (General disorders) | 0 (0) | 4 (5) | 1 (1) | 6 (7) | 7 (7) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 7 (7) | 5 (7) | 5 (6) | 23 (33) | 30 (43) | 3 (4) | 8 (8)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (4) | 1 (1) | 10 (11) | 20 (36) | 4 (9) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (2) | 2 (2) | 8 (12) | 18 (25) | 5 (6) | 3 (3)
Urinary tract infection (Infections and infestations) | 5 (5) | 2 (2) | 2 (2) | 17 (19) | 17 (23) | 8 (8) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 3 (4) | 9 (10) | 13 (18) | 3 (4) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 11 (11) | 14 (17) | 3 (4) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1) | 2 (2) | 12 (13) | 10 (16) | 4 (4) | 2 (2)
Weight decreased (Investigations) | 1 (1) | 4 (5) | 3 (3) | 12 (12) | 17 (17) | 4 (5) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 20 (21) | 8 (10) | 11 (12) | 36 (43) | 51 (55) | 9 (9) | 8 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (9) | 3 (3) | 12 (21) | 11 (21) | 3 (7) | 1 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 4 (5) | 3 (3) | 9 (9) | 8 (10) | 4 (7) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (6) | 3 (3) | 2 (3) | 19 (28) | 10 (11) | 6 (11) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 6 (7) | 7 (9) | 36 (52) | 24 (37) | 9 (13) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 5 (5) | 6 (6) | 24 (31) | 21 (27) | 3 (3) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 1 (1) | 18 (20) | 15 (15) | 4 (5) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 4 (7) | 19 (23) | 14 (15) | 3 (3) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 5 (5) | 18 (25) | 19 (25) | 4 (4) | 1 (4)
Dizziness (Nervous system disorders) | 9 (9) | 4 (4) | 3 (3) | 19 (25) | 18 (27) | 3 (4) | 7 (7)
Headache (Nervous system disorders) | 8 (8) | 9 (11) | 7 (10) | 21 (33) | 30 (45) | 8 (11) | 6 (10)
Anxiety (Psychiatric disorders) | 4 (6) | 4 (4) | 1 (1) | 10 (10) | 8 (8) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 8 (8) | 2 (2) | 3 (3) | 9 (10) | 11 (12) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 13 (13) | 6 (8) | 37 (50) | 42 (50) | 7 (7) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 10 (10) | 1 (1) | 18 (20) | 29 (33) | 7 (7) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 4 (4) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5) | 3 (4) | 4 (4) | 10 (11) | 1 (1) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6) | 4 (4) | 6 (6) | 49 (77) | 57 (74) | 6 (7) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 4 (5) | 3 (3) | 29 (38) | 33 (49) | 11 (15) | 7 (9)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 10 (11) | 18 (23) | 3 (4) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (7) | 11 (11) | 2 (2) | 3 (5)
Leukopenia (Blood and lymphatic system disorders) | 8 (8) | 3 (6) | 4 (7) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 7 (14) | 5 (8) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (12) | 7 (10) | 2 (2) | 3 (5) | 3 (5) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 4 (4) | 2 (3) | 0 (0) | 3 (4) | 7 (7) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 1 (1) | 0 (0) | 4 (8) | 10 (11) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 11 (13) | 9 (10) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 6 (6) | 12 (12) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 9 (11) | 7 (10) | 0 (0) | 0 (0)
Chest pain (General disorders) | 3 (3) | 3 (4) | 1 (1) | 7 (8) | 11 (15) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 3 (3) | 5 (5) | 10 (11) | 11 (13) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 3 (3) | 0 (0) | 7 (9) | 2 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 6 (11) | 2 (5) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 2 (2) | 3 (3) | 5 (9) | 7 (14) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (4) | 3 (4) | 2 (2) | 6 (17) | 7 (8) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 3 (4) | 4 (5) | 2 (10) | 1 (5) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 5 (7) | 4 (9) | 5 (8) | 2 (9) | 5 (9) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 5 (6) | 3 (3) | 3 (3) | 4 (12) | 3 (3) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 3 (7) | 3 (4) | 7 (15) | 6 (7) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 5 (7) | 7 (18) | 10 (25) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (5) | 3 (4) | 2 (2) | 5 (6) | 12 (13) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (10) | 3 (3) | 2 (2) | 8 (8) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6) | 2 (3) | 5 (5) | 9 (11) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4) | 3 (3) | 2 (2) | 8 (8) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 5 (5) | 4 (4) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 6 (6) | 7 (7) | 5 (7) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 3 (3) | 5 (6) | 3 (3) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 4 (4) | 4 (4) | 1 (1) | 7 (7) | 12 (13) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10) | 15 (18) | 11 (11) | 7 (8) | 2 (4) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 18 (24) | 18 (18) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (2) | 10 (12) | 7 (8) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 14 (19) | 16 (19) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 9 (9) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.